CLINICAL TRIAL: NCT01367431
Title: Xanthohumol and Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: Oregon State University (Other)
Collaborators: Oregon Health and Science University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jan Frederik Stevens, Associate Professor of Medicinal Chemistry, Department of Pharmaceutical Sciences, College of Pharmacy, Oregon State University
Other Study IDs: R21AT005294 (NIH); R21AT005294 (NIH)
Record Dates: First submitted 2011-03-15; First posted 2011-06-07 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Metabolic Syndrome
Keywords: Xanthohumol; Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — xanthohumol

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 20 mg: Single dose 20 mg Xanthohumol
  Interventions: Dietary Supplement: Xanthohumol
- 60 mg: Single dose 60 mg Xanthohumol
  Interventions: Dietary Supplement: Xanthohumol
- 180 mg: Single dose 180 mg Xanthohumol
  Interventions: Dietary Supplement: Xanthohumol

INTERVENTIONS:
Dietary Supplement: Xanthohumol — PK study with one capsule of one of the three doses randomly assigned

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (PK) of xanthohumol (XN). Small amounts of xanthohumol occur naturally in hops, used to make beer, and XN is also found in beer itself. Studies in animals have shown that XN can lower blood sugar and blood lipids such as triglycerides, which can contribute to heart disease. The purpose of this study is to see how much of the XN is absorbed into the blood and how fast it leaves the body when taken by mouth. Once the PK study has been done, the investigators' long-term goal is to learn if xanthohumol can lower risk factors for heart disease and type-2 diabetes in humans.

ELIGIBILITY:
* BMI 18-32 kg/m2 (to avoid confounders with extreme obesity).
* Smoking or non-smoking.
* Having normal or clinically acceptable physical examination and clinical laboratory tests.
* Willing to abstain from beer consumption for four days prior to and during the study because beer contains XN and related prenylated (PN) flavonoids, such as IX, 8-PN and 6-PN.
* Not currently taking prescription drugs.
* Not having had acute medical conditions, such as hospitalizations or surgeries, at least three months prior to entry into the study.
* If female, not pregnant (as confirmed by urine pregnancy test), breastfeeding, or planning to become pregnant before completing the study, and using effective method of contraception (hormonal methods NOT permitted).
* If male with a partner of childbearing potential, willing to inform their partner of their participation in this clinical study and use highly effective methods of birth control during the study.
* Not currently following an extreme diet, such as Atkin's, Zone or Ornish, and willing to maintain their current diet without extreme changes for the duration of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women in the Portland, Oregon area
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Levels of xanthohumol and metabolites. | 6 days
  The outcome measures will be the levels of xanthohumol and its metabolites in blood and urine following a single dose of 20 mg, 60mg, or 180 mg of xanthohumol over a course of six days. These levels will be used to determine the pharmacokinetics of xanthohumol in humans.

CONTACTS AND LOCATIONS:
Overall Officials: Jan F Stevens, PhD, Principal Investigator — Oregon State University; Jon Q Purnell, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States